CLINICAL TRIAL: NCT01990651
Title: The Use of Circulating Tumor Cells in Non-Small Cell Lung Cancer: Novel Isolation Methods and Clinical Applications
Brief Title: Study of Use of CTC in NSCLC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Responsible Party: Sponsor
Other Study IDs: 15847
Record Dates: First submitted 2013-11-15; First posted 2013-11-21 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2013-11

CONDITIONS: Non Small Cell Lung Cancer; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to assess whether the detection of circulating tumor cells (CTC) could be used as a tool to earlier diagnose, more accurately predict treatment response / failure and predict overall survival in non-small cell lung cancer (NSCLC) patients

DETAILED DESCRIPTION:
Lung cancer remains the most common cause of cancer mortality in the world for both men and women. More than half of patients diagnosed will die within the first year. Given these concerning facts, we are in need of novel methodologies to diagnose patients at earlier stages of the disease, more accurately predict treatment response / failure and predict overall survival.

The use of CTC has been investigated and shown to predict progression free survival and overall survival in metastatic breast cancer, and recommended as a breast cancer tumor marker by the American Society of Clinical Oncology. There have also been relationships between CTC's and survival, shown in metastatic colorectal and prostate cancer. However, CTC's have not been thoroughly investigated in non-small cell lung cancer. This trial will assess if the detection of circulating tumor cells could be used as a tool to help further advance treatment for NSCLC patients.

ELIGIBILITY:
Inclusion Criteria:

For subjects with lung malignancies:

* 18 years of age and older
* Diagnosis of new or recurrent non-small cell lung cancer
* Awaiting treatment and follow up
* Have radiographic measurable metastatic disease that can be followed
* Be able to sign an IRB approved informed consent form
* Life expectancy greater than 12 weeks

For subjects with COPD and without lung malignancies:

* 18 years of age and older
* Diagnosis of COPD
* No current or prior malignancies (except squamous or basal cell carcinoma of the skin)
* Be able to sign an IRB approved informed consent form

For Healthy Control Subjects (Dry Runs):

* 18 years of age and older
* Has no current or prior malignancies (except squamous or basal cell carcinoma of the skin)
* Patients must sign an IRB approved informed consent form

Exclusion Criteria:

For subjects with lung malignancies:

* Have other concurrent lung cancer malignancies, or any other form of malignancy (except squamous or basal cell carcinoma of the skin)
* ECOG performance status of 4
* Pregnant female (self-reporting)
* Cognitively Impaired
* Prisoner

For subjects with COPD and without lung malignancies and Healthy Controls:

* Any other form of malignancy (except squamous or basal cell carcinoma of the skin)
* Pregnant female (self reporting)
* Cognitively impaired
* Prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2011-09; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
To estimate the correlation between the number of circulating tumor cells (CTC) and clinical stage of the disease | Completed within 6 months of the last sample collected
In Stage I, II or III patients with resectable disease, to obtain preliminary data to assess whether the number of CTC in post operative peripheral blood samples decrease compared with the number of CTC in the pre operative peripheral blood samples | Measured up to 12 week post op
To obtain preliminary data to assess whether lower numbers of CTC are associated with a reduction in tumor burden (by RECIST criteria) on imaging | Completed within 6 months of the last sample collected
To obtain preliminary data to assess whether there is a decrease in the number of CTC during treatment with chemotherapy in Stage IV disease | measured up to completion of 4 cycles of chemo or up to 12 weeks after completion of radiation and chemo treatment

SECONDARY OUTCOMES:
To obtain preliminary data on the association of baseline number of CTC and disease-free survival for patients with all stages of disease | Will be assessed for up to 2 years after subjects last visit
To obtain preliminary data on the association of baseline number of CTC and overall survival for patients with all stages of disease | Will be assessed for up to 2 years after subjects last visit

CONTACTS AND LOCATIONS:
Overall Officials: Thao Dang, MD, Principal Investigator — University of Virginia Health System
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States